CLINICAL TRIAL: NCT03311490
Title: A Randomized Pilot Trial to Evaluate the Preliminary Effect and Safety of Using Spraino® to Prevent Lateral Ankle Sprains in Indoor Sports (The Spraino Pilot Trial)
Brief Title: The Spraino Pilot Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision to halt the trial in October was made in June, as the anticipated no. of events(ankle sprains) required for the analyses was almost reached in June
Sponsor: Spraino (Industry)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Aalborg University (Other); Metropolitan University College (Other); The Copenhagen Center for Health Technology (CACHET) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4559
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Athletes With Previous Lateral Ankle Sprain(s)
Keywords: Ankle Sprain; Prophylaxis; Indoor Sports; Ligamentous sprain; Prevention
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants allocated to the intervention group will use Spraino® as a measure to prevent lateral ankle sprains.
  Interventions: Device: Spraino
- Control (No Intervention): Participants allocated to the control group will be a "do-as-usual" comparator. This implies, that the participants can treat and prevent lateral ankle sprains in any way they wish, except using Spraino®.

INTERVENTIONS:
Device: Spraino — Participants allocated to the intervention group will use Spraino® as a measure to prevent future lateral ankle sprains during all on-court practice sessions and matches. Spraino® is an adhesive polytetrafluoroethylene (PTFE or "Teflon") patch. It is developed with the intent of minimizing lateral shoe- surface friction whenever initial contact is carried out in an inverted position of the ankle joint. Each Spraino® PTFE patch has a minimum durability of 20 hours use and will be provided by the trial sponsor, Spraino® ApS. The participants allocated to the intervention group will receive four pairs of the Spraino® patches via postal service or by hand delivery on a monthly basis, or upon request if material is worn out prematurely during the 52-week trial period.
  Arms: Intervention

SUMMARY:
This pilot study will establish the preliminary effect and safety of using Spraino® to prevent lateral ankle sprains amongst athletes competing in indoor sports at sub-elite level, with a one-year follow-up.

All recruited participants will have a history of lateral ankle sprain in the preceding 24 months prior to the initiation of the trial. Half of the included participants will receive Spraino® to prevent lateral ankle sprains (intervention group). The other half will receive no intervention ("do-as-usual" control group). Both groups will be permitted to continue or initiate any usual care of their choice, except Spraino® in the control group. Short Message Services (SMS) will be used for registration of injury and exposure.

DETAILED DESCRIPTION:
The purpose of this exploratory trial (named "The Spraino Pilot Trial") is to establish the preliminary effect and safety of using Spraino® to prevent lateral ankle sprains amongst athletes competing in indoor sports at sub-elite level (handball, basketball, floorball and badminton) when compared to a "do-as-usual" control group.

It is a randomized controlled pilot trial (Pilot-RCT) with a two-group parallel design and blinded outcome assessment. The trial will include prospective injury and exposure registration using a Short Message Services-system (SMS-Track) throughout a 52-week follow-up period (one calendar year).

It is anticipated that 500 participants, which approximates to 250 in each group, will be enrolled in the trial. The enrollment process will cease when at least 250 participants have been allocated to the intervention group. Only athletes participating in indoor sports with a history of a lateral ankle sprain in the preceding 24 months are eligible for inclusion in the trial. The participants will be randomized (1:1 allocation ratio) using numbered lots. The randomization process will ensure stratification for gender, sports discipline and level of play.

A full trial protocol, based on the "SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials" (Chan et al., 2013) and the "PREPARE Trial guide" (Bandholm et al., 2017), will be published and made publicly available. The trial report will adhere to the CONSORT 2010 statement, using the extension for randomized pilot and feasibility trials.

Being an exploratory pilot trial, the study is designed with a flat outcome structure with multiple evenly valued outcome measures. Thus, no primary and secondary outcome measure hierarchy exists.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 years old at commencement of trial.
* Participant can read, speak and understand Danish.
* Participant can receive and reply to texts on a cell phone using Short Message Services (SMS).
* Participant performs indoor sports (Handball, basketball, floorball orbadminton) in a sub-elite level team with ≥ 2 weekly practice sessions.
* Participant has incurred ≥ 1 lateral ankle sprain injury in the preceding 24 months.
* Participant has returned to play at commencement of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Lateral ankle sprains | 52 weeks
  Rate of lateral ankle sprains (continuous)
  The incidence rate is defined as the number of lateral ankle sprains per 1000 hours of exposure.
First-time non-contact lateral ankle sprains | 52 weeks
  Rate of first-time non-contact lateral ankle sprains (continuous)
  The incidence rate is defined as the number of first-time non-contact lateral ankle sprains per 1000 hours of exposure.
Time-loss due to first-time non-contact lateral ankle sprains | 52 weeks
  Time-loss (in number of weeks) due to first-time non-contact lateral ankle sprains per athlete (continuous)
Severe first-time non-contact lateral ankle sprains | 52 weeks
  Rate of severe first-time non-contact lateral ankle sprains (continuous)
  The incidence rate is defined as the number of severe first-time non-contact lateral ankle sprains (≥ 3 weeks with time-loss) per 1000 hours of exposure.
Recurrent non-contact lateral ankle sprains | 52 weeks
  Rate of recurrent non-contact lateral ankle sprains (continuous)
  The incidence rate is defined as the number of recurrent non-contact lateral ankle sprains per 1000 hours of exposure.
Time-loss due to recurrent non-contact lateral ankle sprains | 52 weeks
  Time-loss (in number of weeks) due to recurrent non-contact lateral ankle sprains per athlete (continuous)
Severe recurrent non-contact lateral ankle sprains | 52 weeks
  Rate of severe recurrent non-contact lateral ankle sprains (continuous)
  The incidence rate is defined as the number of severe recurrent non-contact lateral ankle sprains (≥ 3 weeks with time-loss) per 1000 hours of exposure.
First-time lateral ankle sprains | 52 weeks
  Rate of first-time lateral ankle sprains (continuous)
  The incidence rate is defined as the summation of both contact and non-contact first-time lateral ankle sprains per 1000 hours of exposure.
Time-loss due to first-time lateral ankle sprains | 52 weeks
  Time-loss (in number of weeks) due to first-time lateral ankle sprains per athlete (continuous)
Severe first-time lateral ankle sprains | 52 weeks
  Rate of severe first-time lateral ankle sprains (continuous)
  The incidence rate is defined as the number of severe first-time lateral ankle sprains (≥ 3 weeks with time-loss) per 1000 hours of exposure.
Recurrent lateral ankle sprains | 52 weeks
  Rate of recurrent lateral ankle sprains (continuous)
  The incidence rate is defined as the summation of both contact and non-contact recurrent lateral ankle sprains per 1000 hours of exposure.
Time-loss due to recurrent lateral ankle sprains | 52 weeks
  Time-loss (in number of weeks) due to recurrent lateral ankle sprains per athlete (continuous)
Severe recurrent lateral ankle sprains | 52 weeks
  Rate of severe recurrent lateral ankle sprains (continuous)
  The incidence rate is defined as the number of severe recurrent lateral ankle sprains (≥ 3 weeks with time-loss) per 1000 hours of exposure.

OTHER OUTCOMES:
Adverse effects from using Spraino® | 52 weeks
  Reports of adverse events in the intervention group (binary)
  All adverse events will be registered while the participants are enrolled in the trial. Adverse events will be reported as type and number of events. The included participants will be encouraged to report any adverse events related to the use of Spraino® to the trial hotline.
Fear of re-injury | 52 weeks
  Fear of lateral ankle sprain re-injury (continuous)
  Change in fear of re-injury from pre- to post-trial intervention period. Fear of re-injury is scored on a numeric rating scale from 0 - 100 (0 = Extremely fear full, 100 = No fear at all)
Ankle pain | 52 weeks
  Ankle pain (continuous)
  Change in ankle pain from pre- to post-trial intervention period. Ankle pain is scored on a numeric rating scale from 0 - 10 (0 = No pain at all, 10 = Extremely painful)

CONTACTS AND LOCATIONS:
Overall Officials: Filip G Lysdal, MSc, Principal Investigator — Center for Sensory Motor Interaction, Department of Health Science and Technology, Aalborg University, Denmark; Kristian Thorborg, PhD, Study Director — Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C), Clinical Research Centre, Amager-Hvidovre Hospital, Copenhagen University, Hvidovre, Denmark; Thomas Q Bandholm, PhD, Study Chair — Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C), Clinical Research Centre, Amager-Hvidovre Hospital, Copenhagen University, Hvidovre, Denmark; Eamonn Delahunt, PhD, Study Chair — School of Public Health, Physiotherapy and Sports Science, University College Dublin, Dublin, Ireland
Locations (2):
- Denmark (2):
  - Physical Activity and Human Performance, Center for Sensory Motor Interaction, Department of Health Science and Technology, Aalborg University, Denmark, Aalborg
  - Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C), Clinical Research Centre, Amager-Hvidovre Hospital, Copenhagen University, Hvidovre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Bandholm T, Christensen R, Thorborg K, Treweek S, Henriksen M. Preparing for what the reporting checklists will not tell you: the PREPARE Trial guide for planning clinical research to avoid research waste. Br J Sports Med. 2017 Oct;51(20):1494-1501. doi: 10.1136/bjsports-2017-097527. Epub 2017 Sep 7. No abstract available. PMID 28882839
- [Derived] Lysdal FG, Bandholm T, Tolstrup JS, Clausen MB, Mann S, Petersen PB, Gronlykke TB, Kersting UG, Delahunt E, Thorborg K. Does the Spraino low-friction shoe patch prevent lateral ankle sprain injury in indoor sports? A pilot randomised controlled trial with 510 participants with previous ankle injuries. Br J Sports Med. 2021 Jan;55(2):92-98. doi: 10.1136/bjsports-2019-101767. Epub 2020 Aug 12. PMID 32796016
- See also: SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. — https://doi.org/10.1136/bmj.e7586
- See also: Preparing for what the reporting checklists will not tell you: the PREPARE Trial guide for planning clinical research to avoid research waste. — http://dx.doi.org/10.1136/bjsports-2017-097527